CLINICAL TRIAL: NCT06707402
Title: The Effects of 24 Weeks Community-based Brisk Walking on Physical Function, Comorbidities, Cognition, Disease Severity, and Health-related Quality of Life in People With Parkinson's Disease.
Brief Title: The Effects of 24-Weeks Community-based Brisk Walking in People With Parkinson's Disease
Acronym: We-Walk-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Karolinska Institutet (Other); Viborg Regional Hospital (Other); Danish Parkinson Association (Other); Fonden af 2. Juli 1984 til bekÃ¦mpelse af Parkinsons Sygdom, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Walking and PD
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Brisk walking; Walking difficulty
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combined individual home-based and supervised group-based walking exercise (Experimental): 43 people with Parkinsons disease would be randomly assigned to this experimental group. The group will receive the intervention "WALK", that covers a personalized exercise program and group exercise session. It further covers the same as in the HOME group.
  Interventions: Behavioral: WALK
- Individual home-based exercise (Active Comparator): 43 people with Parkinsons disease would be randomly assigned to this active comparator group. The group receives the intervention (HOME) that covers an activity tracker and motivational telephone calls. It further covers the same as in the CON group.
  Interventions: Behavioral: ACTIVE
- Control group (Sham Comparator): 43 people with Parkinsons disease would be randomly assigned to this sham comparator group. The group will only receive a short lecture in Parkinsons disease and exercise after completing the baseline test and allocated to the group.
  Interventions: Behavioral: CON

INTERVENTIONS:
Behavioral: WALK — The intervention covers a personalized 24-week progressive brisk walking program. The program consists of moderate to high-intensity walking (i.e., 55-85% maximal heart rate) performed as both continuous and interval training sessions 2-3 times/week lasting 30-60 min/session. Four individually supervised sessions will be conducted in the first 2 weeks, while 1 supervised group session will be received bi-weekly. Furthermore, the group will receive an activity tracker and monthly telephone calls will be offered to adjust the intensity of the program (if necessary), clarify any questions regarding the intervention, and give verbal motivation. At the baseline assessment and at week 12, during a group training session, the figure of 8 walk test will be conducted to gain insigh tinto the current status of the training program. Lastly, after completion of the baseline test, the participants are given a brief educational session (walking advice) on recommended guidelines for physical activity
  Arms: Combined individual home-based and supervised group-based walking exercise
Behavioral: ACTIVE — Will receive an activity tracker is provided alongside monthly telephone calls and walking advice after the baseline test. Similar to WALK, 3 telephone calls are provided during the follow-up period.
  Arms: Individual home-based exercise
Behavioral: CON — Receives a brief educational session (walking advice) is provided at baseline, after which no further contacts are made.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate if brisk walking can improve walking function in people with Parkinson's disease and what kind of brisk walking intervention that is most effective. The main questions are:

If brisk walking can reduce self-perceived walking difficulty What type of exercise intervention is most effective. Researchers will compare a brisk walking group receiving a personalized walking program with a group receiving an activity tracker and a control group.

Participants will

* be tested at baseline (0 weeks), post the intervention period (24 weeks) and after a follow-up period (48 weeks).
* be randomly allocated to one of three groups at baseline.
* follow the prescribed intervention they are allocated to.

DETAILED DESCRIPTION:
Background Parkinson's disease is a progressive neurodegenerative disorder and one of the leading causes of disability worldwide. Impaired walking is considered one of the most bothersome symptoms that people with Parkinson's disease wish to improve, affecting independence, ability to work, and quality of life. Walking impairment is present from the early stage of the disease with an expected progression and a more frequent presentation along the course of the disease. Currently, only few medical treatments exist that target walking, and these show minor effects while causing side effects. Non-pharmacological interventions that can improve or prevent loss of walking ability are therefore highly warranted.

Exercise is a promising non-pharmacological intervention in people with Parkinson's disease with studies reporting improved walking performance following different exercise modalities, including high-intensity aerobic exercise. Despite extensive research investigating the effects of various exercise interventions on walking, few have examined more traditional walking training. This is somewhat surprising as walking is task-specific training for walking itself, while also being feasible and showing promising results in people with Parkinson's disease. In addition, walking is easily accessible and a potential efficient low-cost intervention that is commonly used and therefore well-known in clinical rehabilitation practice. Yet only two long-term studies could be located applying walking training. Despite being long-term, these studies are limited by 1) not considering possible factors facilitating adherence, 2) not performing follow-up testing, 3) not applying any inclusion criterion for walking impairment implying that any potential effects might be diminished due to well-functioning participants without walking impairments, 4) not including a comprehensive test battery (i.e., no registration of comorbidities, physical activity level, health-related quality of life), and 5) not investigating the effect on perceived walking difficulties despite the relevance of understanding the subjective impact of walking training. Further evaluation of walking interventions is therefore needed in people with Parkinson's disease.

Despite the importance of a physically active lifestyle, only 27% (potentially less) of people with Parkinson's disease meet the established physical activity recommendations (≥ 150 min/week of moderate to vigorous physical activity). Therefore, it is very challenging to design a walking intervention that increases physical activity levels while being sustainable. To do so, it is essential to incorporate motivational factors that facilitate adherence. These include high self-efficacy, low cost, less travel, self-perceived positive effects of walking, and support from family/carers and health professionals. To comply with these factors, remotely or partly supervised home-based exercise has been suggested as a feasible and effective strategy to alleviate Parkinson's disease motor symptoms. Another aspect to consider is group vs. individually based exercise sessions. Both have shown equally effective in improving functional capacity in healthy individuals, but combined group- and individual-based exercise has been recommended as the most attractive model for the broadest range of people with Parkinson's disease. Overall, by incorporating these strategies in walking training, this exercise modality might offer a sustainable, cost-effective, and easy-to-apply intervention that can be offered in local communities worldwide. This would also include people with Parkinson's disease living without easy access to training facilities or who are governed by poor healthcare systems. Another even more easy-to-apply and low-cost intervention to increase physical activity, is to offer a wearable activity tracker. One study reported increased physical activity level in people with Multiple sclerosis when offering a wearable activity tracker and engaging in group- and individual motivational online meetings compared to a control group. However, to the investigator's knowledge, this has not been assessed in people with Parkinson's disease.

Therefore, the primary aim is to investigate the efficacy of a 24-week combined supervised group- and non-supervised individual-based walking intervention (WALK) compared to both a group receiving a wearable activity tracker (HOME) and a control group (CON) on perceived walking difficulties in people with Parkinson's disease. The secondary aims are to identify and characterize responders and non-responders to walking training and to investigate the cost-effectiveness of these exercise interventions.

The hypothesis is that the WALK group will be superior to HOME and CON, while HOME will be superior to CON after 24 weeks in reducing perceived walking difficulties, which will be sustained after a 24-week follow up.

Methods and materials The project includes one main study and two embedded studies. Study 1 (main study): A single-blinded randomized controlled trial including three interventions (WALK, HOME and CON). Tests will be conducted at 0, 24 and 48 weeks.

Study 2: Identification and characterization of responders (i.e., ≥3 point decrease in the generic walking scale or ≥6% increase in maximal oxygen consumption) and non-responders to walking training.

Study 3: Economic evaluation of WALK compared to HOME and CON.

Statistical considerations The study sample size is powered based on descriptive Parkinson's disease data on the primary outcome (i.e., generic walking scale) and the assumption that a clinically meaningful change of ≥3 points will be detected between all three groups after 24 weeks (i.e. WALK > HOME > CON). Moreover, based on the inclusion criteria, a more homogeneous population sample compared to the previous study is expected, and thus a lower standard deviation. Lastly, it is expected that 15% will drop out. A one-way ANOVA was used to estimate the sample size (a=0.05, power=0.8, 24-weeks post mean values for CON, HOME and WALK = 15, 12, 9 ± 8, and dropout proportion = 15%). The calculation showed that 43 people with Parkinson's disease should be enrolled into each group.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed with Parkinson's disease
2. aged ≥40 years
3. Hoehn and Yahr stage ≤3
4. able to independently undertake transportation back and forth from test days and training sessions
5. expectedly able to complete ≥85% of the training sessions
6. experience walking difficulties (the generic walking scale (Walk-12G) score ≥8.5).

Exclusion Criteria:

1. have another neurological disorder or other disorders that affect gait and balance (e.g., severe arthritis or arthrosis)
2. are pregnant
3. have dementia (Montreal Cognitive Assessment score <18)
4. are suffering from alcohol abuse (i.e., exceeding ten units per week, according to the Danish Health Authority recommendation
5. have cardiovascular, respiratory, orthopedic, or metabolic disorders or other medical comorbidities hindering participation in maximal exercise testing.
6. have a depression
7. use an activity tracker during exercise
8. performing high-intensity brisk walking three or more times during a week.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender
Enrollment: 129 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The Generic Walking Scale - 12 items (Walk-12G) | From enrollment to the end of follow-up at 48 weeks
  The generic walking scale is a 12-item questionnaire covering different aspects of walking difficulties during everyday life. Scores ranged from 0 (no problem) to 42 (severe walking difficulties)

SECONDARY OUTCOMES:
Demographic measures | From enrollment to the end of follow-up at 48 weeks
  Demographic measures cover the following:
  Sex (male/female) Age (years) Weight (kg) Height (cm) Body mass index (kg/m2) Fat mass (%) Muscle mass (kg) Time of diagnosis (years) Blood pressure (mmHg) Years of education (years) Levodopa Equivalent Daily Dose (Parkinson's disease medication) Beta blocker (yes/no)
Chair rise | From enrollment to the end of follow-up at 48 weeks
  Linear encoder equipment is used to measure muscle force and muscle power during a chair rise.
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating scale (MDS-UPDRS) part I, II, III, and IV | From enrollment to the end of follow-up at 48 weeks
  All four parts (I to IV) are collected during the study as well as the individual motor symptoms from part III (rigidity, bradykinesia, postural instability and tremor) Part I assesses non-motor symptoms experience of daily life. Score ranged from 0 (no problem) to 52 (severe problems) Part II assesses motor symptoms experienced of daily life. Score ranged from 0 (no problem) to 52 (severe problems) Part III is a motor examination. Scores ranged from 0 (no problem) to 132 (severe problems) Part IV assesses motor complications. Scores ranged from 0 (no problem) to 24 (severe problems) Rigidity covers items 3.3 and scores from 0 (no problem) to 20 (severe problems). Bradykinesia covers items 3.4-3.8 and 3.14 and scores from 0 (no problem) to 44 (severe problems) postural instability covers items 3.9-3.13 and scores from 0 (no problem) to 20 (severe problems). Tremor covers items 3.15-3.18 and scores from 0 (no problem) to 40 (severe problems).
Mini Balance Evaluation Systems Test (MiniBESTest) | From enrollment to the end of follow-up at 48 weeks
  Assess balance. Scores from 0 (worse) to 28 (best) points
Timed-up and Go (TUG) | From enrollment to the end of follow-up at 48 weeks
  Three trials are performed. The fastest trial is used for analysis.
Six-Spot Step Test (SSST) | From enrollment to the end of follow-up at 48 weeks
  Four trials are performed (two for right leg and two for left leg). The average time for the four trials are used in the analysis
Six-minute walk test (6MWT) | From enrollment to the end of follow-up at 48 weeks
  Total distance (m) covered during 6 minutes of fast walking
The Montreal Cognitive Assessment (MoCA) test | From enrollment to the end of follow-up at 48 weeks
  Scores from 0 (worse) to 30 (best). Total score are used in the analysis
Symbol Digit Modalities Test (SDMT) | From enrollment to the end of follow-up at 48 weeks
  Measures cognition. Test duration is 90 sec. Score of 0 is worse, and the higher the better. There is no limit but often not more than 75 points.
Maximal oxygen consumption test (VO2max test) | From enrollment to the end of follow-up at 48 weeks
  Maximal oxygen consumption test (VO2max) would be performed on a ergometer bicycle. VO2max (O2 ml/min) will be measured. Weight would be used to calculate weight normalized VO2max (O2 ml/kg/min)
Borg scale (part of VO2max test) | From enrollment to the end of follow-up at 48 weeks
  The Borg scale assesses self-perceived exertion. It ranges from 6 (minor exertion) to 20 (maximum exertion). The scale would be used as part of the VO2max test.
Maximal heart rate (part of VO2max test) | From enrollment to the end of follow-up at 48 weeks
  Maximal heart rate (beats/min) would be obtained as part of the VO2max test. The highest measure would be used for further analysis.
Physcial activity level | From enrollment to the end of follow-up at 48 weeks
  Physical activity level will be assessed using accelerometer (Axivity A3) for 7 consecutive days.
Physical Activity Enjoyment Scale (PACES) (questionnaire) | Only at the post test (24 weeks)
  The short version with 8 items will be used for both interventions groups (WALK and ACTIVE). It assesses the enjoyment of performing physical activity and scores ranged from 0 (no enjoyment) to 56 (greatest level of enjoyment)
Baecke Physical Activity Questionnaire (BHPAQ) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess physical activity during work and leisure time and amount of sport participation. Scores ranged from 1 (low activity) to 5 (a lot of activity) in the three categories.
EuroQol-5 Domain-5 level (EQ-5D-5L) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess quality of life. Scores in Denmark ranged from -0.757 (worse quality of life) to 1.0 (best quality of life).
Modfied Fatigue Impact Scale (MFIS) (questionnaire) | Baseline only
  The questionnaire are included to be used in future cross-sectional analyses. It assesses fatigue and scores ranged from 0 (not fatigue) to 84 (extremely fatigued). The questionnaire is also subdivided into physical (0-36 points) cognitive (0-40 points) and psychosocial (0-8 points) subscales.
Major Depression Inventory (MDI) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  It assesses depression symptoms. Scores ranged from 0 (no depression) to 50 (severe depression)
Non-Motor Symptoms Questionnaire (NMSQuest) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess non-motor symptoms and contains 30 items. It scores from 0 (no symptoms) to 30 (severe symptoms)
Parkinsons Disease Questionnaire-39 items (PDQ-39) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess quality of life. It is specific for Parkinsons disease. It contains several domains. The total score ranged from 0 (no problem) to 100 (severe problems).
Parkinsons disease Fatigue Scale-16 items (PFS-16) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Parkinson specific survey that assesses fatigue. Score ranged from 16 (no fatigue) and 80 (severe fatigue)
The Pittsburgh Sleep Quality Index (PSQI) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess sleep quality. Contains 10 items (and some additional items). Score ranged from 0 (no problem) to 21 (severe problem)
Breif Pain Inventory (BPI) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess pain and interference. It contains 16 items, and the score is divided in pain which goes from 0 (no pain) to 40 (worst pain) and interference of pain which goes from 0 (no interference) to 70 (extreme interference).
Falls Efficacy Scale - International (FES-I) (questionnaire) | From enrollment to the end of follow-up at 48 weeks
  Assess fear of falling. Contains 16 items. Score ranged from 16 (no fear) to 64 (severe fear)

OTHER OUTCOMES:
Figure-of-8 Walk Test (F8W) | Baseline and midway through the intervention (12 weeks)
  The F8W is included to motivate participants in the WALK group to sustain active. The test would be conducted at baseline (after randomization) and midway through the intervention period (12 weeks). By seeing progress (i.e., improved test performance) the participant would be motivated to sustain active. Otherwise, if no improvement is detected, the training program would be reevaluated for the participant to increase the likelihood of an improved walking function (i.e., improved Walk-12G score) after 24 weeks.
Motivational telephone calls | From enrollment to the end of follow-up at 48 weeks
  Both WALK and ACTIVE will receive motivational telephone calls. By the end of the call, three questions (yes/no answer) would be asked to the participants to assess the degree of motivation through the intervention period and follow-up period. In total 8 telephone calls would be conducted (5 during the intervention period and 3 during the follow-up period)
  The questions are:
  1. Du you feel motivated to continuing the training in the following period?
  2. Have you felt that the training gave you more energy during the day?
  3. Do you feel that you have made progress with your training in the latest period?
  4. Do you feel that the training has improved your general health and wellbeing?

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department of Public Health, Sport Science, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make the individual data available for other researchers. This requires informed consents from each participant and a data processing agreement, according to the GDPR rules, which have not been prepared prior to the initiation of the study. However, a co-supervisor (Erika Franzén, Sweden) affiliated to the project might receive some relevant pseudonymized data. If that is the case, the protocol description will be updated.

REFERENCES:
- [Background] Lindh-Rengifo M, Jonasson SB, Ullen S, Mattsson-Carlgren N, Nilsson MH. Perceived walking difficulties in Parkinson's disease - predictors and changes over time. BMC Geriatr. 2021 Apr 1;21(1):221. doi: 10.1186/s12877-021-02113-0. PMID 33794786
- [Background] Frost R, Levati S, McClurg D, Brady M, Williams B. What Adherence Measures Should Be Used in Trials of Home-Based Rehabilitation Interventions? A Systematic Review of the Validity, Reliability, and Acceptability of Measures. Arch Phys Med Rehabil. 2017 Jun;98(6):1241-1256.e45. doi: 10.1016/j.apmr.2016.08.482. Epub 2016 Oct 1. PMID 27702555
- [Background] Rudmik L, Drummond M. Health economic evaluation: important principles and methodology. Laryngoscope. 2013 Jun;123(6):1341-7. doi: 10.1002/lary.23943. Epub 2013 Mar 11. PMID 23483522
- [Background] Chaudhuri KR, Martinez-Martin P, Brown RG, Sethi K, Stocchi F, Odin P, Ondo W, Abe K, Macphee G, Macmahon D, Barone P, Rabey M, Forbes A, Breen K, Tluk S, Naidu Y, Olanow W, Williams AJ, Thomas S, Rye D, Tsuboi Y, Hand A, Schapira AH. The metric properties of a novel non-motor symptoms scale for Parkinson's disease: Results from an international pilot study. Mov Disord. 2007 Oct 15;22(13):1901-11. doi: 10.1002/mds.21596. PMID 17674410
- [Background] Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. Am J Clin Nutr. 1982 Nov;36(5):936-42. doi: 10.1093/ajcn/36.5.936. PMID 7137077
- [Background] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Background] Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4. doi: 10.1007/pl00007730. PMID 9617716
- [Background] Pascoe M, Alamri Y, Dalrymple-Alford J, Anderson T, MacAskill M. The Symbol-Digit Modalities Test in Mild Cognitive Impairment: Evidence from Parkinson's Disease Patients. Eur Neurol. 2018;79(3-4):206-210. doi: 10.1159/000485669. Epub 2018 Mar 29. PMID 29597229
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Clarke CL, Taylor J, Crighton LJ, Goodbrand JA, McMurdo MET, Witham MD. Validation of the AX3 triaxial accelerometer in older functionally impaired people. Aging Clin Exp Res. 2017 Jun;29(3):451-457. doi: 10.1007/s40520-016-0604-8. Epub 2016 Jul 19. PMID 27435918
- [Background] Bonde-Jensen F, Dalgas U, Hvid LG, Langeskov-Christensen M. Validity and reliability of linear encoder muscle power testing in persons with Parkinson's disease. Clin Rehabil. 2024 May;38(5):678-687. doi: 10.1177/02692155231224987. Epub 2024 Jan 9. PMID 38193269
- [Background] Brincks J, Callesen J, Johnsen E, Dalgas U. A study of the validity of the Six-Spot Step Test in ambulatory people with Parkinson's disease. Clin Rehabil. 2019 Jul;33(7):1206-1213. doi: 10.1177/0269215519833016. Epub 2019 Feb 25. PMID 30798635
- [Background] Brincks J, Callesen J, Dalgas U, Johnsen E. Test-retest reliability and limits of agreement of the Six-Spot Step Test in people with Parkinson's disease. Clin Rehabil. 2019 Feb;33(2):285-292. doi: 10.1177/0269215518803144. PMID 30789075
- [Background] Morris S, Morris ME, Iansek R. Reliability of measurements obtained with the Timed "Up & Go" test in people with Parkinson disease. Phys Ther. 2001 Feb;81(2):810-8. doi: 10.1093/ptj/81.2.810. PMID 11175678
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Hoops S, Nazem S, Siderowf AD, Duda JE, Xie SX, Stern MB, Weintraub D. Validity of the MoCA and MMSE in the detection of MCI and dementia in Parkinson disease. Neurology. 2009 Nov 24;73(21):1738-45. doi: 10.1212/WNL.0b013e3181c34b47. PMID 19933974
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Soke F, Erkoc Ataoglu NE, Ozcan Gulsen E, Yilmaz O, Gulsen C, Kocer B, Kirteke F, Basturk S, Comoglu SS, Tokcaer AB. The psychometric properties of the figure-of-eight walk test in people with Parkinson's disease. Disabil Rehabil. 2023 Jan;45(2):301-309. doi: 10.1080/09638288.2022.2028020. Epub 2022 Feb 22. PMID 35191344
- [Background] Lowry K, Woods T, Malone A, Krajek A, Smiley A, Van Swearingen J. The Figure-of-8 Walk Test used to detect the loss of motor skill in walking among persons with Parkinson's disease. Physiother Theory Pract. 2022 Apr;38(4):552-560. doi: 10.1080/09593985.2020.1774948. Epub 2020 Jun 16. PMID 32543340
- [Background] Jensen FB, Dalgas U, Brincks J, Langeskov-Christensen M. Validity and reliability of VO2-max testing in persons with Parkinson's disease. Parkinsonism Relat Disord. 2023 Apr;109:105324. doi: 10.1016/j.parkreldis.2023.105324. Epub 2023 Feb 15. PMID 36827950
- [Background] Bladh S, Nilsson MH, Hariz GM, Westergren A, Hobart J, Hagell P. Psychometric performance of a generic walking scale (Walk-12G) in multiple sclerosis and Parkinson's disease. J Neurol. 2012 Apr;259(4):729-38. doi: 10.1007/s00415-011-6254-z. Epub 2011 Sep 29. PMID 21956376
- [Background] Plow M, Finlayson M, Liu J, Motl RW, Bethoux F, Sattar A. Randomized Controlled Trial of a Telephone-Delivered Physical Activity and Fatigue Self-management Interventions in Adults With Multiple Sclerosis. Arch Phys Med Rehabil. 2019 Nov;100(11):2006-2014. doi: 10.1016/j.apmr.2019.04.022. Epub 2019 Jun 21. PMID 31229528
- [Background] Larsen RT, Wagner V, Korfitsen CB, Keller C, Juhl CB, Langberg H, Christensen J. Effectiveness of physical activity monitors in adults: systematic review and meta-analysis. BMJ. 2022 Jan 26;376:e068047. doi: 10.1136/bmj-2021-068047. PMID 35082116
- [Background] Ferguson T, Olds T, Curtis R, Blake H, Crozier AJ, Dankiw K, Dumuid D, Kasai D, O'Connor E, Virgara R, Maher C. Effectiveness of wearable activity trackers to increase physical activity and improve health: a systematic review of systematic reviews and meta-analyses. Lancet Digit Health. 2022 Aug;4(8):e615-e626. doi: 10.1016/S2589-7500(22)00111-X. PMID 35868813
- [Background] King AC, Haskell WL, Taylor CB, Kraemer HC, DeBusk RF. Group- vs home-based exercise training in healthy older men and women. A community-based clinical trial. JAMA. 1991 Sep 18;266(11):1535-42. PMID 1880885
- [Background] Flynn A, Dennis S, Preston E, Canning CG, Allen NE. Exercising with Parkinson's: The good, the bad and the need for support to keep exercising. A qualitative study. Clin Rehabil. 2022 Oct;36(10):1332-1341. doi: 10.1177/02692155221100884. Epub 2022 May 13. PMID 35549564
- [Background] Girnis JL, Cavanaugh JT, Baker TC, Duncan RP, Fulford D, LaValley MP, Lawrence M, Nordahl T, Porciuncula F, Rawson KS, Saint-Hilaire M, Thomas CA, Zajac JA, Earhart GM, Ellis TD. Natural Walking Intensity in Persons With Parkinson Disease. J Neurol Phys Ther. 2023 Jul 1;47(3):146-154. doi: 10.1097/NPT.0000000000000440. Epub 2023 Apr 4. PMID 37016469
- [Background] Benka Wallen M, Franzen E, Nero H, Hagstromer M. Levels and Patterns of Physical Activity and Sedentary Behavior in Elderly People With Mild to Moderate Parkinson Disease. Phys Ther. 2015 Aug;95(8):1135-41. doi: 10.2522/ptj.20140374. Epub 2015 Feb 5. PMID 25655884
- [Background] Reuter I, Mehnert S, Leone P, Kaps M, Oechsner M, Engelhardt M. Effects of a flexibility and relaxation programme, walking, and nordic walking on Parkinson's disease. J Aging Res. 2011;2011:232473. doi: 10.4061/2011/232473. Epub 2011 Mar 30. PMID 21603199
- [Background] Paul SS, Canning CG, Lofgren N, Sherrington C, Lee DC, Bampton J, Howard K. People with Parkinson's disease are more willing to do additional exercise if the exercise program has specific attributes: a discrete choice experiment. J Physiother. 2021 Jan;67(1):49-55. doi: 10.1016/j.jphys.2020.12.007. Epub 2020 Dec 24. PMID 33358546
- [Background] Hornby TG, Rafferty MR, Pinto D, French D, Jordan N. Cost-Effectiveness of High-intensity Training vs Conventional Therapy for Individuals With Subacute Stroke. Arch Phys Med Rehabil. 2022 Jul;103(7S):S197-S204. doi: 10.1016/j.apmr.2021.05.017. Epub 2021 Jul 3. PMID 34228956
- [Background] Robinson AG, Dennett AM, Snowdon DA. Treadmill training may be an effective form of task-specific training for improving mobility in people with Parkinson's disease and multiple sclerosis: a systematic review and meta-analysis. Physiotherapy. 2019 Jun;105(2):174-186. doi: 10.1016/j.physio.2018.11.007. Epub 2018 Nov 15. PMID 30876717
- [Background] Mak MKY, Wong-Yu ISK. Six-Month Community-Based Brisk Walking and Balance Exercise Alleviates Motor Symptoms and Promotes Functions in People with Parkinson's Disease: A Randomized Controlled Trial. J Parkinsons Dis. 2021;11(3):1431-1441. doi: 10.3233/JPD-202503. PMID 33967056
- [Background] Gamborg M, Hvid LG, Dalgas U, Langeskov-Christensen M. Parkinson's disease and intensive exercise therapy - An updated systematic review and meta-analysis. Acta Neurol Scand. 2022 May;145(5):504-528. doi: 10.1111/ane.13579. Epub 2022 Jan 8. PMID 34997759
- [Background] Wilson J, Alcock L, Yarnall AJ, Lord S, Lawson RA, Morris R, Taylor JP, Burn DJ, Rochester L, Galna B. Gait Progression Over 6 Years in Parkinson's Disease: Effects of Age, Medication, and Pathology. Front Aging Neurosci. 2020 Oct 15;12:577435. doi: 10.3389/fnagi.2020.577435. eCollection 2020. PMID 33192470
- [Background] Port RJ, Rumsby M, Brown G, Harrison IF, Amjad A, Bale CJ. People with Parkinson's Disease: What Symptoms Do They Most Want to Improve and How Does This Change with Disease Duration? J Parkinsons Dis. 2021;11(2):715-724. doi: 10.3233/JPD-202346. PMID 33459664
- [Background] Koerts J, Konig M, Tucha L, Tucha O. Working capacity of patients with Parkinson's disease - A systematic review. Parkinsonism Relat Disord. 2016 Jun;27:9-24. doi: 10.1016/j.parkreldis.2016.03.017. Epub 2016 Mar 22. PMID 27029582
- [Background] Mirelman A, Bonato P, Camicioli R, Ellis TD, Giladi N, Hamilton JL, Hass CJ, Hausdorff JM, Pelosin E, Almeida QJ. Gait impairments in Parkinson's disease. Lancet Neurol. 2019 Jul;18(7):697-708. doi: 10.1016/S1474-4422(19)30044-4. Epub 2019 Apr 8. PMID 30975519
- [Background] Uebelacker LA, Epstein-Lubow G, Lewis T, Broughton MK, Friedman JH. A survey of Parkinson's disease patients: most bothersome symptoms and coping preferences. J Parkinsons Dis. 2014;4(4):717-23. doi: 10.3233/JPD-140446. PMID 25271239
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468